CLINICAL TRIAL: NCT03258177
Title: Utilization of Virtual Care in Postoperative Patients to Improve the Patient Experience
Brief Title: Virtual Visits (Utilization of Virtual Care in Postoperative Patients to Improve the Patient Experience)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American College of Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00082477; 07-17-14E (Other: Atrium)
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2021-09

CONDITIONS: Appendectomy, Laparoscopic; Cholecystectomy, Laparoscopic; Cholecystectomy, Robotic
Keywords: Virtual Visits; Telehealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Visit Group (Experimental): Participants assigned to the virtual visit group will receive a virtual visit as their postoperative follow-up visit.
  Interventions: Other: Virtual Visit
- Standard In-person Group (No Intervention): Participants assigned to the standard in-person group will receive an in-person follow-up visit as their postoperative follow-up visit.

INTERVENTIONS:
Other: Virtual Visit — Participants will be given information about how to enroll in virtual care. Participants will use their own camera-enabled device with internet connection to see and speak to the medical professional in real-time and complete the virtual follow-up visit.
  Arms: Virtual Visit Group

SUMMARY:
The purpose of this study is to implement and evaluate postoperative virtual care visits for patients who undergo a laparoscopic appendectomy, laparoscopic cholecystectomy, or robotic cholecystectomy. The investigators aim to better understand whether postoperative virtual care visits will not result in a greater composite measure of the occurrence of hospital encounters within Atrium Health (AH) for the 30 days following surgery than standard in-person clinic care. The investigators also aim to better understand whether postoperative virtual care visits provide time and cost savings, and provide equal or improved patient satisfaction and convenience.

DETAILED DESCRIPTION:
Participants will be randomized to complete either a postoperative follow-up visit using virtual care technology or by attending a standard in-person visit at the clinic. The virtual visit uses a camera-enabled device and internet access to provide live access to the medical professional. Surveys to assess patient satisfaction and convenience will be administered by email on the day of the postoperative follow-up visit. Additional information including demographics, hospital encounters within 30 days of surgery, length of time of the follow-up visit, travel cost and time, whether additional follow-up care is required, and complications after surgery will be collected to evaluate postoperative virtual care visits. Subject participation in the study will end after follow-up care is complete or at 30 days, whichever occurs last.

ELIGIBILITY:
Inclusion Criteria:

* Willing to comply with all study procedures and be available for the duration of the study
* English speaking
* Able to read
* Have an email address
* Scheduled to undergo a laparoscopic appendectomy, laparoscopic cholecystectomy or robotic cholecystectomy OR have undergone an unplanned (urgent or emergent) laparoscopic appendectomy, laparoscopic cholecystectomy, or robotic cholecystectomy
* Have surgery performed by a surgeon at either Carolinas Medical Center-Main or Carolinas Medical Center- Mercy who provides emergency general surgery clinical coverage
* Live in North Carolina or South Carolina

Exclusion Criteria:

* Unable to complete a virtual visit (due to lack of appropriate technology, necessary technology skills, other);
* Medical condition, laboratory finding, or physical exam finding that precludes participation (patients at high risk for complications, particularly those with perforated appendicitis, patients with active cocaine abuse)
* Postoperative length of stay greater than or equal to 4 days
* Discharged with drains that need to be removed at a postoperative visit
* Admitted from or discharged to assisted living facility, skilled nursing facility, or location other than home
* Have chronic pain for which the participant takes narcotic medication

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Composite measure of the occurrence of hospital encounters | from date of surgery until the date of 30 days after surgery
  composite measure of the occurrence of hospital encounters for the 30 days following surgery including all-cause and any-site inpatient, observational, and emergency department visits within Carolinas HealthCare System

SECONDARY OUTCOMES:
Postoperative follow-up visit time length in minutes | date of follow-up visit, approximately 14 days after date of surgery
  total time of postoperative follow-up visit in minutes
Patient satisfaction score | date of follow-up visit, approximately 14 days after date of surgery
  self-reported patient satisfaction rating for follow-up visit assessed by survey
Patient convenience score | date of follow-up visit, approximately 14 days after date of surgery
  self-reported patient convenience rating for follow-up visit assessed by survey
Rate of postoperative follow-up | date of follow-up visit, approximately 14 days after date of surgery
  percent of patients who receive a postoperative follow-up visit
Rate of postoperative no-shows | date of follow-up visit, approximately 14 days after date of surgery
  percent of scheduled postoperative follow-up appointments in which patients do not complete
Patient travel time to clinic in minutes | date of follow-up visit, approximately 14 days after date of surgery
  total patient travel time from home to postoperative follow-up clinic in minutes
Patient cost savings in dollars | date of follow-up visit, approximately 14 days after date of surgery
  Patient gas cost savings for travel from home to postoperative follow-up clinic

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Reinke, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harkey K, Connor CD, Wang H, Kaiser N, Matthews BD, Kelz R, Reinke CE. View from the Patient Perspective: Mixed-Methods Analysis of Post-Discharge Virtual Visits in a Randomized Controlled Trial. J Am Coll Surg. 2021 Nov;233(5):593-605.e4. doi: 10.1016/j.jamcollsurg.2021.07.688. Epub 2021 Sep 9. PMID 34509613
- [Derived] Harkey K, Kaiser N, Zhao J, Hetherington T, Gutnik B, Matthews BD, Kelz RR, Reinke CE. Postdischarge Virtual Visits for Low-risk Surgeries: A Randomized Noninferiority Clinical Trial. JAMA Surg. 2021 Mar 1;156(3):221-228. doi: 10.1001/jamasurg.2020.6265. PMID 33439221

DOCUMENTS (1):
  • Informed Consent Form (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT03258177/ICF_000.pdf